CLINICAL TRIAL: NCT03974841
Title: Cornual Wedge Resection for Interstitial Pregnancy and Postoperative Outcome
Brief Title: Cornual Wedge Resection Outcome
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019.06
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Ectopic Pregnancy; Laparoscopic; Cornual Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic; Pregnancy, Cornual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic cornual resection — patients undergoing laparoscopic cornual resection due to cornual ectopic pregnancy

SUMMARY:
Cornual pregnancy is a rare form of ectopic pregnancy that accounts for 2% to 4% of ectopic pregnancies, with a mortality rate between 2.0% and 2.5%. Traditionally, interstitial pregnancies were treated by laparotomy with cornial resection or hysterectomy. However, nowadays, increasingly interstitial pregnancies are treated by laparoscopic cranial resection.

Although this technique can potentially protect the fertility of the patient, it carries a serious risk of bleeding and requires a surgical experience.

ELIGIBILITY:
Inclusion Criteria:

* cornual ectopic pregnancy
* Patients undergoing laparoscopic cornual wedge resection

Exclusion Criteria:

* medical treatment area due to cornual pregnancy
* laparotomy
* conservatively managed patients

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: postoperative results of patients who underwent laparoscopic cornual resection for cornual ectopic pregnancy, Patients forming the study group will be operated in the center for the last 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Operation time | surgery from start to end
  The duration of surgery of patients undergoing laparoscopic cornual resection due to cornual ectopic pregnancy
amount of bleeding | 48 hours
  The amount of hemorrhage in patients undergoing laparoscopic cornual resection due to cornual ectopic pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)